CLINICAL TRIAL: NCT05770648
Title: A Prospective, Multicenter, Randomized Controlled Trial to Evaluate the Efficacy and Safety of the Transcatheter Tricuspid Valvuloplasty System in Patients With Severe or Above Tricuspid Regurgitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Huihe Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSP-K-02
Record Dates: First submitted 2023-03-05; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- K-clipTM transcatheter annuloplasty system+Guideline Directed Medical Therapy GDMT (Experimental)
  Interventions: Device: Transcatheter Annuloplasty
- Guideline Directed Medical Therapy, GDMT (Other)
  Interventions: Other: The guidelines guide medication

INTERVENTIONS:
Device: Transcatheter Annuloplasty — Under the guidance of ultrasound, the transcatheter tricuspid ring forming system accurately reaches the designated position of the tricuspid valve region through the jugular vein and superior vena cava approach. The expanded tricuspid ring tissue is clammed together with the clamping parts and anchor parts, and the circumference of the tricuspid ring is reduced, thus reducing the area of the opening of the tricuspid valve that cannot be closed originally, and achieving the purpose of minimally invasive treatment of tricuspid regurgitation.
  Arms: K-clipTM transcatheter annuloplasty system+Guideline Directed Medical Therapy GDMT
Other: The guidelines guide medication — The guidelines guide medication
  Arms: Guideline Directed Medical Therapy, GDMT

SUMMARY:
To evaluate the efficacy and safety of the transcatheter tricuspid valve ring system produced by Shanghai Huihe Medical Technology Co., Ltd. in the treatment of patients with severe or above tricuspid regurgitation who cannot be evaluated by clinicians for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥60, male or female; (2) Patients with severe or above secondary tricuspid regurgitation (TR≥4+) (secondary tricuspid regurgitation: tricuspid regurgitation caused by right atrial disease, right ventricular cardiomyopathy, right ventricular myocardial infarction, left heart valve disease, congenital heart disease and other diseases); (3) A multidisciplinary cardiac team consisting of cardiovascular physicians, cardiovascular surgeons, imaging physicians, anesthesiologists, and at least 2 physicians considered the subjects to be at high risk for surgical procedures, i.e., EuroScore II was greater than 3.0%; (4) Left ventricular ejection fraction LVEF≥30%; (5) The subject voluntarily participates in the clinical trial and agrees or his guardian agrees to sign the informed consent; (6) Symptoms of tricuspid regurgitation, such as chest tightness, asthma, shortness of breath, lower limb edema, ascites; (7) NYHA Grades 2 to 4, including Grades 2 and 4; (8) The optimal drug treatment for tricuspid valve ≥ 30 days and the patient's state was stable; (9) Patients with mitral regurgitation, atrial fibrillation, coronary artery disease, and heart failure should be treated for ≥ 30 days with medication or ≥ 30 days after instrument therapy and in stable condition.

Exclusion Criteria:

1. Patients with pure organic (i.e. primary) tricuspid regurgitation;
2. Patients with pulmonary artery systolic blood pressure ≥60 mmHg;
3. Patients with tricuspid valve prosthesis or plastic ring, or patients with tricuspid valve-related surgery;
4. Patients with retrotricuspid annulus calcification;
5. Evidence of intracardiac, jugular and superior vena cava masses, thrombus or growths;
6. Patients with more than moderate aortic stenosis, mitral stenosis, aortic regurgitation, or mitral regurgitation;
7. Patients with severe uncontrolled hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg);
8. Percutaneous coronary intervention within 1 month;
9. Myocardial infarction or known unstable angina within the previous 1 month;
10. cerebrovascular accidents occurred within the previous 3 months;
11. Patients with active endocarditis or active rheumatic heart disease;
12. Patients with coagulopathy, hypercoagulability or anemia (hemoglobin < 90 g/L);
13. Patients in the acute infection stage or other severe infections;
14. Patients with active peptic ulcer or active gastrointestinal bleeding;
15. severe end-stage diseases (such as malignant tumors, severe lung diseases, liver diseases, renal failure) with a life expectancy of less than 1 year;
16. Patients with known allergy or contraindications to the raw material or drug (e.g. antiplatelet drugs, anticoagulants) of the test product;
17. persons addicted to alcohol, drugs or drugs;
18. Patients with cognitive impairment;
19. A history of epilepsy or mental illness with primary and persistent seizures and poor drug control;
20. Participate in any other clinical trial (other than a registered study) within 30 days prior to signing the informed consent;
21. have had a pacemaker (other than a leadless pacemaker) or a defibrillator implanted in the past, or plan to have a pacemaker (other than a leadless pacemaker) or a defibrillator implanted;
22. tricuspid stenosis;
23. Ebstain syndrome;
24. esophageal esophageal echocardiography (TEE) and Trans thoracic echocardiography (TTE) were not esophageal esophageal tricuspid ring anatomy;
25. Hemodynamic instability;
26. Patients with chronic dialysis;
27. Women who have planned to become pregnant during pregnancy, lactation or clinical study;
28. Other conditions for which the investigator considers it inappropriate to participate in the clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects with no all-cause death, no heart failure readmitted, NYHA increased by one grade or more, and TR decreased ≥1+ within 6 months after randomization. | Within 6 months of randomization
  The percentage of subjects with no all-cause death, no heart failure readmitted, NYHA increased by one grade or more, and TR decreased ≥1+ within 6 months after randomization.